CLINICAL TRIAL: NCT00186225
Title: Stem Cell Transplantation From Matched Unrelated or Partially Matched Related Donors Using a Preparatory Regimen Consisting of Fractionated Total Body Irradiation (FTBI) and Cyclophosphamide (CY)
Brief Title: Stem Cell Transplant From Matched Unrelated or Partially Matched Related Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13390; 75268 (Other: Old IRB number); BMT22 (Other: OnCore)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Blood Cancer; Blood and Marrow Transplant (BMT)
MeSH Terms: conditions — Hematologic Neoplasms

INTERVENTIONS:
Procedure: ablative allogeneic hematopoietic cell transplantation

SUMMARY:
To evaluate the use of unrelated donors for hematopoietic cell transplantation in the treatment of hematologic and lymphoid malignancies.

DETAILED DESCRIPTION:
Stem Cell Transplantation from Matched Unrelated or Partially Matched Related Donors Using a Preparatory Regimen Consisting of Fractionated Total Body Irradiation (FTBI) and Cyclophosphamide (CY). To administer high dose radio-chemotherapy followed by stem cell transplantation from a matched unrelated donor or a partially matched related donor.

ELIGIBILITY:
Inclusion Criteria:- acute leukemia

* chronic leukemia
* lymphoblastic lymphoma
* MDS
* MPS Exclusion Criteria:- organ dysfunction
* HIV positive

Ages: 4 Weeks to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 1989-11; Primary Completion 2007-06 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
oxicity and efficacy of TBI and cyclophosphamide as preparation for hematopoietic cell transplantation from partially matched and unrelated donors.

SECONDARY OUTCOMES:
Overall Survival
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnston, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States